CLINICAL TRIAL: NCT07236437
Title: Living Well Program: Impact on Healthcare Costs and Clinical Outcomes in Breast Cancer Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scott A. Irwin, MD, PhD (Other)
Collaborators: Prosoma (Unknown); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor-Investigator, Scott A. Irwin, MD, PhD, Principal Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2024-12-Irwin-LivingWell
Record Dates: First submitted 2025-10-30; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Supportive Care in Cancer; Depression
Keywords: Anxiety; Breast Cancer; Telecoaching; Telehealth; Supportive Care
MeSH Terms: conditions — Anxiety Disorders; Depression; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study has one, non-randomized treatment arm. The second arm is retrospectively matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Arm (Experimental): The intervention arm will participate in the Living Well app modules and telecoaching sessions.
  Interventions: Device: Living Well Program

INTERVENTIONS:
Device: Living Well Program — The intervention is multicomponent, including a mobile application and telecoaching. The mobile application is comprised of 21 modules integrating psychoeducation and cognitive-behavioral therapy principles, designed to be completed in 3 months. Modules require 15-30 minutes to complete and address topics such as breast cancer education, anxiety management, and adaptive coping strategies. Telecoaching services will provide personalized support for cancer patients throughout their treatment. Participants will complete five 20-30 minute telecoaching sessions with qualified mental health professionals over 6 months.
  Outcomes will be compared to a retrospective control cohort.

SUMMARY:
The goal of this study is to evaluate the efficacy and cost-effectiveness of the Living Well Program, a digital therapeutic application with telecoaching support, in breast cancer patients with moderate-to-severe anxiety. The main question the study aims to answer is: does digital cognitive-behavioral therapy-based interventions decrease the overall healthcare costs of patients with stage II to IV breast cancer?

The study has one group of participants who will use the Living Well app and telecoaching support. This group will be compared to retroactively matched controls. Over 3 months, patients will complete 21 mental health modules and 5 telecoaching sessions. In the following 3 months, they will complete any outstanding telecoaching sessions and modules while still being monitored, even if they finished all modules and sessions in the first 3 months. The 6 months after that will be the follow-up phase. They will still have access to the Living Well app and may continue to use it, and they will complete the same assessment questionnaires as baseline to identify any changes in their overall mental health.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, historically controlled interventional study. It will evaluate the effectiveness and healthcare impacts of a digital cognitive-behavioral therapy-based intervention for anxiety in patients with stage II to IV breast cancer. The high prevalence of anxiety among cancer patients with limited access to mental health support drives higher total healthcare costs, healthcare services utilization, and worse clinical outcomes. This is one of the major rationales for the study. There have been promising preliminary results from previous studies of this intervention in reducing anxiety and depression in cancer patients.

There are minimal known potential risk: primarily, the potential for psychological distress associated with responding to questions about health status and employment. Known potential benefits to patients in the intervention group include immediate psychological well-being improvements and decreased anxiety associated with breast cancer diagnosis and treatment. Long term, patients may develop improved coping and emotional regulations skills that persist beyond the study period. These skills may enhance quality of life and improve treatment adherence and outcomes. More broadly, this study may offer societal benefits through an improved understanding of digital therapeutic interventions in oncology care. Economic analyses from this study may provide insights to the cost-effectiveness of digital interventions in healthcare.

This trial utilizes retrospectively matched controls based on key demographic and clinical characteristics as a comparison group to the intervention group.

Use of retrospectively matched controls was chosen due to the nature of the intervention and the target population. Given that the Living Well Program is a digital therapeutic intervention aimed at addressing a significant unmet need in cancer care, it was deemed ethically preferable to offer the intervention to all eligible participants rather than withholding it from a control group.

The intervention consists of 21 modules in the mobile application, and five 20-minute telecoaching sessions. Participants begin with the first module upon enrollment and are asked to complete one module every other day, or as needed, with each module taking 15-30 minutes. This regimen is designed to be completed over a 6-month period, constituting the planned maximum dosage. The 15-30-minute module duration aims to provide meaningful engagement without overburdening patients undergoing cancer treatment. The 3-month active intervention period aligns with typical durations of effective cognitive-behavioral therapy interventions, while extended 12-month access to the application allows for continued support and skill reinforcement. The inclusion of five telecoaching sessions for the first six months provides human support to complement the digital intervention, an approach shown to enhance engagement and outcomes in digital mental health interventions.

The baseline assessment will include comprehensive demographic and medical history questionnaire, treatment history and sociodemographic factors. Patients will complete validated psychometric scales to assess their quality of life and mental health, including the Generalized Anxiety Disorder-7 (GAD-7) to measure anxiety symptoms, Patient Health Questionnaire-9 (PHQ-9) to measure depression symptoms, PROMIS-29 to assess quality of life, and the Edmonton Symptom Assessment System (ESAS) to assess physical symptoms. They will also complete the Cedars-Sinai Wellbeing Screen and 10-Point Distress thermometer. These assessments provide baseline measures of participants overall mental health.

The intervention will be administered through a smartphone app called The Living Well Program. A study team member will assist with installation and configuration of the app so patients can complete modules and engage in telecoaching sessions. Follow-up assessments at 3-, 6-, and 12-months post-baseline will include the same questionnaires as the baseline assessment, collection of healthcare costs and utilization from medical records, assessment of concomitant medications, and evaluation of intervention adherence and engagement metrics from the app.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. First time breast cancer diagnosis
3. Established with a Cedars-Sinai Surgical or Medical Oncologist for cancer care and is within 30 days of starting or having started adjuvant or neoadjuvant therapy
4. Prognosis of greater than 1 year
5. Breast cancer staging of II-IV
6. Moderate to severe anxiety (GAD-7 >= 10)
7. English language proficiency
8. Smartphone and ability to use the application as assessed by study staff (IG only)
9. Signed dated informed consent form (ICF) within 30 days of diagnosis (IG only)

Exclusion Criteria:

1. Prior history of different cancer diagnosis or recurrence of the same cancer
2. Serious mental illness evidenced by patient self-report, chart review and/or diagnosis codes
3. Presence of suicidal ideation as measured by the Ask Suicide-Screening Questions (ASQ) or a history of suicide attempts as evidenced by self-report or chart review
4. Current active addiction (drugs, alcohol, etc.) evidenced by Opioid Risk Tool, chart review and/or diagnosis codes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Study participants total healthcare costs from enrollment to six months compared to controls. | From baseline assessment to 6-month time point.
  Healthcare costs will be extracted from electronic medical records. "Healthcare Costs" will include a sum of the costs of the following over a six month timeframe (enrollment to six months): emergency department visits, ICU visits, inpatient hospital charges, unscheduled hospitalizations, hospital days above expected, 30-day readmissions, outpatient visits, diagnostic visits, medications, chemotherapy, immunotherapy, targeted therapies, pathology, imaging, radiation, and any other treatments.

SECONDARY OUTCOMES:
Study participants total healthcare costs from baseline to 3-months compared to controls. | From baseline to 3-month time point.
  Healthcare costs will be extracted from patient's electronic medical records from baseline assessment to three months. They will be compared to controls over the same period.
  "Healthcare Costs" will include the cost of the following: emergency department visits, ICU visits, inpatient hospital charges, unscheduled hospitalizations, hospital days above expected, 30-day readmissions, outpatient visits, diagnostic visits, medications, chemotherapy, immunotherapy, targeted therapies, pathology, imaging, radiation, and any other treatments.
Study participants total number of healthcare utilization events from baseline to 3-months compared to controls. | From baseline assessment to 3-month time point.
  Healthcare utilization will be extracted from CS-Link EMR for participants and controls over the same time period. Assessment of utilization measures the number of the following events:
  * Emergency department (ED) visits
  * Intensive Care Unit (ICU) visits
  * Inpatient hospital charges
  * Unscheduled hospitalizations
  * Hospital days above expected
  * 30-day readmissions
  * Outpatient visits
  * Diagnostic visits
  * Medications, chemotherapy, immunotherapy, targeted therapies, pathology, imaging, radiation, and other treatments
  Healthcare utilization score will be the total number of healthcare utilization events in the given time period (e.g., 1 emergency department visit and 1 unscheduled hospitalization = healthcare utilization score of 2).
Changes in study participant's anxiety scores from baseline to 3 months. | From baseline to 3 months time point.
  Changes will be measured using the Generalized Anxiety Disorder-7 (GAD-7) assessment for anxiety. Participant's GAD-7 assessment scores at baseline will be compared to GAD-7 score at 3-months time point. A higher GAD-7 score indicates more severe anxiety.
Study participants total healthcare costs from baseline to 12-months compared to controls. | From baseline to 12-month time point.
  Healthcare costs will be extracted from patient's electronic medical records from baseline assessment to 12 months. They will be compared to controls over the same period.
  "Healthcare Costs" will include the cost of the following: emergency department visits, ICU visits, inpatient hospital charges, unscheduled hospitalizations, hospital days above expected, 30-day readmissions, outpatient visits, diagnostic visits, medications, chemotherapy, immunotherapy, targeted therapies, pathology, imaging, radiation, and any other treatments.
Study participants total number of healthcare utilization events from baseline to 6-months compared to controls. | From baseline to 6-month time point.
  Healthcare utilization will be extracted from CS-Link EMR for participants and controls over the same time period. Assessment of utilization measures the number of the following events:
  * Emergency department (ED) visits
  * Intensive Care Unit (ICU) visits
  * Inpatient hospital charges
  * Unscheduled hospitalizations
  * Hospital days above expected
  * 30-day readmissions
  * Outpatient visits
  * Diagnostic visits
  * Medications, chemotherapy, immunotherapy, targeted therapies, pathology, imaging, radiation, and other treatments
  Healthcare utilization score will be the total number of healthcare utilization events in the given time period (e.g., 1 emergency department visit and 1 unscheduled hospitalization = healthcare utilization score of 2).
Study participants total number of healthcare utilization events from baseline to 12-months compared to controls. | From baseline to 12-month time point.
  Healthcare utilization will be extracted from CS-Link EMR for participants and controls over the same time period. Assessment of utilization measures the number of the following events:
  * Emergency department (ED) visits
  * Intensive Care Unit (ICU) visits
  * Inpatient hospital charges
  * Unscheduled hospitalizations
  * Hospital days above expected
  * 30-day readmissions
  * Outpatient visits
  * Diagnostic visits
  * Medications, chemotherapy, immunotherapy, targeted therapies, pathology, imaging, radiation, and other treatments
  Healthcare utilization score will be the total number of healthcare utilization events in the given time period (e.g., 1 emergency department visit and 1 unscheduled hospitalization = healthcare utilization score of 2).
Changes to participant's anxiety score from baseline to 6-months. | From baseline to 6-months time point.
  Changes will be measured using the Generalized Anxiety Disorderr-7 (GAD-7) assessment for anxiety. Participant's GAD-7 assessment scores at baseline will be compared to GAD-7 score at 6-months time point. A higher GAD-7 score indicates more severe anxiety.
Changes to study participant's anxiety scores from baseline to 12-months. | From baseline to 12- months time point.
  Changes will be measured using the Generalized Anxiety Disorder-7 (GAD-7) assessment for anxiety. Participant's GAD-7 assessment scores at baseline will be compared to GAD-7 score at 12-months time point. A higher GAD-7 score indicates more severe anxiety.
Study participants changes in depression score from baseline to 3 months. | From baseline to 3-months time point.
  Changes will be measured using the Patient Health Questionnaire-9 (PHQ-9) assessment for depression. Participant's PHQ-9 assessment scores at baseline will be compared to PHQ-9 score at 3-months time point. A higher PHQ-9 score indicates more severe depression symptoms.
Study participants depression score changes from baseline to 6-months. | From baseline to 6-months time point.
  Changes will be measured using the Patient Health Questionnaire-9 (PHQ-9) assessment for depression. Participant's PHQ-9 assessment scores at baseline will be compared to PHQ-9 score at 6-months time point. A higher PHQ-9 score indicates more severe depression symptoms.
Study participants depression score changes over 12- months. | From baseline to 12-months time point.
  Changes will be measured using the Patient Health Questionnaire-9 (PHQ-9) assessment for depression. Participant's PHQ-9 assessment scores at baseline will be compared to PHQ-9 score at 12-months time point. A higher PHQ-9 score indicates more severe depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Irwin, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No